CLINICAL TRIAL: NCT05317000
Title: A Window Trial of 5-Azacytidine or Nivolumab or Combination Nivolumab Plus 5-Azacytidine in Resectable HPV-Associated Head and Neck Squamous Cell Cancer
Brief Title: 5-Azacytidine and/or Nivolumab in Resectable HPV-Associated HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Burtness (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor-Investigator, Barbara Burtness, Professor of Medicine, Medical Oncology, Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000025632; 1P50DE030707-01 (NIH)
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: HPV- Associated Head and Neck Squamous Cell Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Azacitidine

STUDY DESIGN:
Intervention Model Description: This Phase 2 study is a 3-arm window trial, randomizing patients to pre-operative treatment with 5-azacytidine alone, to nivolumab alone, or the combination of 5-azacytidine and nivolumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: 5-azacytidine (Active Comparator): Patients will receive 5-azacytidine 75mg/m2 IV daily x 5. Treatment must begin on a Monday.
  Patients will receive anti-emetic premedication with prochlorperazine 10 mg IV, a 5HT3 antagonist per institutional guidelines, aprepitant or fos-aprepitant, and prn lorazepam on day 1. Day 2-5 patients will receive prochlorperazine 10 mg IV. Subsequent day 5HT3 antagonist therapy will be determined per institutional guidelines, as recommendations vary based on the half-life of the agent chosen. PRN lorazepam can be used days 2-5.
  Dexamethasone will be reserved for patients who are not controlled by the initial regimen.
  A single cycle of 5-azacytidine will be administered and the patient scheduled for surgery in the period of day 16 through day 18.
  Interventions: Drug: 5-azacytidine
- Arm B: Nivolumab (Active Comparator): Nivolumab will be administered at a dose of 240 mg IV day 1 and day 15. Treatment must be given on a Monday or Tuesday.
  No premedication will be given. Patients will be observed following the initial dose of nivolumab per institutional Surgery will be scheduled in the period of day 16 through day 18.
  Interventions: Drug: Nivolumab
- Arm C: Combination 5-azacytidine and Nivolumab (Experimental): Patients will receive 5-azacytidine 75mg/m2 IV daily x 5. Treatment must begin on a Monday. 5-azacytidine will be given prior to nivolumab on day 2.
  Patients will receive anti-emetic premedication with prochlorperazine 10 mg IV, a 5HT3 antagonist per institutional guidelines, aprepitant or fos-aprepitant, and prn lorazepam on day 1. Day 2-5 patients will receive prochlorperazine 10 mg IV. Subsequent day 5HT3 antagonist therapy will be determined per institutional guidelines, as recommendations vary based on the half-life of the agent chosen. PRN lorazepam can be used days 2-5.
  Nivolumab will be administered at a dose of 240 mg IV day 2 and day 16. No additional premedication will be given on day 16. Dexamethasone will be reserved for patients whose nausea and/or emesis is not controlled by the initial regimen. Surgery will be scheduled in the period of day 17 through day 18.
  Interventions: Drug: Combination 5-azacytidine and nivolumab

INTERVENTIONS:
Drug: Combination 5-azacytidine and nivolumab — The primary objective of the study is to determine whether exposure to the demethylating agent 5-azacytidine will sensitize HPV-associated oropharynx cancer to nivolumab by induction of interferon response, neoantigen expression, and augmentation of lymphocyte infiltration of the tumor microenvironment.
  Other Names: Vidaza and Opdivo
  Arms: Arm C: Combination 5-azacytidine and Nivolumab
Drug: 5-azacytidine — Chemotherapy is the use of drugs to destroy cancer cells. It usually works by keeping the cancer cells from growing, dividing, and making more cells. Because cancer cells usually grow and divide faster than normal cells, chemotherapy has more of an effect on cancer cells. 5-azacytidine works by slowing down the growth of cancer cells. 5-azacytidine has been demonstrated to improve the cell's ability to make some proteins which signal to the immune system.
  Other Names: Vidaza
  Arms: Arm A: 5-azacytidine
Drug: Nivolumab — Immunotherapy is a type of treatment that uses your body's own immune system to help fight cancer. Specifically, Nivolumab belongs to a class of anti-cancer drugs known as immune checkpoint inhibitors. Cancer cells are able to "turn off" the immune system by increasing the production of a protein called PD-1. Nivolumab can block PD-1 and may be able to re-activate the immune response to kill head and neck cancer cells.
  Other Names: Opdivo
  Arms: Arm B: Nivolumab

SUMMARY:
This study is being done because both 5-azacytidine and nivolumab can influence the immune system's response to HPV-associated head and neck cancer, and we wish to evaluate whether taking 5-azacytidine will make HPV-associated head and neck cancer more sensitive to treatment with nivolumab.

5-Azacytidine (5-AZA) is a chemotherapy, and nivolumab is an immunotherapy. Both drugs are approved for use in the US by the Food and Drug Administration (FDA) for use in the treatment of different types of cancer, and nivolumab is approved for use in head and neck cancer that has previously been treated with chemotherapy. Because they are not approved to be used together in HPV-associated head and neck cancer, these drugs are considered experimental in this study. For this study, the drugs will be used either together or separately.

DETAILED DESCRIPTION:
This Phase 2 study is a 3-arm window trial, randomizing patients to pre-operative treatment with 5-azacytidine alone, to nivolumab alone, or the combination of 5-azacytidine and nivolumab. The primary endpoint is immune-related pathologic response, employing the quantitative immune-related pathologic response criteria (ir-PRC) of Cottrell et al. The secondary endpoint is augmentation of tumor infiltration of the tumor microenvironment as determined by a quantitative immunofluorescence score (QIF) measuring CD3+ lymphocytes and granzyme B expression. Secondary endpoints are objective response by modified RECIST, change in Ki-67, change in caspase activity, toxicity and hyperprogression. Patients are eligible with T1-3, N0-2, M0 p16-positive squamous cell carcinoma of the oropharynx deemed resectable by a surgical co-investigator. Patients must have normal absolute lymphocyte count, adequate end organ function, and not require full dose anticoagulation. Patients must be capable of providing, and provide, written informed consent. Patients on Arm A receive 5-azacytidine 75mg/m2 IV once daily day 1-5. Patients on Arm B receive nivolumab 240 mg IV days 1 and 15. Patients on Arm C receive 5-azacytidine as described above and receive nivolumab 240 mg IV days 2 and 16. On arms A and B surgery is performed during the period of days 16 to 18, and on Arm C during the period of days 17 to 18. The study will enroll 8 patients to 5-azacytidine monotherapy and 20 patients per arm to nivolumab or 5-azacytidine/nivolumab combination and has an 80% power to detect a significant difference in immune-related pathologic response, according to the criteria of Cottrell, between the combination arm and each of the monotherapy arms considered separately, using a one-sided Fisher's exact test at a significance level of 0.10.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resectable histologically or cytologically confirmed squamous cell carcinoma of the oropharynx.
2. T1-T3, N0-N2, M0 stage by AJCC 8th edition for HPV-initiated oropharynx cancer.
3. Resectability confirmed by a surgical co-investigator; evaluation may include operative endoscopy to discover second primaries and map tumor extent with biopsy
4. In addition to diagnostic biopsies, biopsies in clinic or at the time of operative endoscopy are required to yield primary tumor for research purposes equivalent to or greater than 3mm cup forceps biopsies X 3. Prior biopsies for research obtained with informed consent for the Yale Biosample Repository Protocol are acceptable if they meet the volume requirements above.
5. HPV-association confirmed by institutional p16 testing (CINtec antibody demonstrating strong and diffuse nuclear and cytoplasmic staining in at least 70% of tumor cells).
6. Age > or equal to 18 years. 5-azacytidine and nivolumab are tolerated in the elderly and there is no upper age limit for patients with adequate performance status.
7. Males and females are eligible.
8. ECOG performance status 0 or 1.
9. Absolute neutrophil count (ANC) > or equal to 1500/microliter, absolute lymphocyte count (ALC) > or equal to 1000/microliter, hemoglobin > or equal to 9 g/dl, platelets > or equal to 100,000/microliter.
10. AST and ALT < 2.5 x upper limit of normal. Bilirubin < 1.5 x upper limit of normal.
11. Albumin > or equal to 3.0 g/dl.
12. Creatinine < or equal to 1.5 x upper limit of normal.
13. Women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study treatment. An extension up to 72 hours prior to the start of study treatment is permissible in situations where results cannot be obtained within the standard 24-hour window.
14. Willing and able to provide written informed consent. Informed consent is required prior to research-related activities, including biopsy. However, if written informed consent for participation in the biosample repository protocol has been obtained, tissue obtained under that consent can be used to meet eligibility criterion 4.

Exclusion Criteria:

1. Medical contraindication to transoral surgery.
2. Full dose anticoagulation.
3. Concomitant invasive malignancy, or malignancy within 2 years except for hormonally responsive breast or prostate cancer, resected non-melanoma skin cancer, resected uterine cervical carcinoma or meningioma.
4. Inability to give informed consent.
5. Prior systemic therapy, radiation, or gross resection for the tumor under study.
6. Women may not be pregnant or breast-feeding.
7. Patients with active autoimmune disease, supraphysiologic systemic corticosteroid use within 7 days, and/or allergies/contraindications to the study drugs are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Increased response for combination therapy compared with either monotherapy | Day 16-18
  As assessed by the ir-PRC of Cottrell.

SECONDARY OUTCOMES:
Increased activated T cell infiltration in 5-Aza containing arms compared to Nivolumab monotherapy arm | Day 16-18
  As confirmed by quantitative immunofluorescence for CD3+ cells and granzyme B expression.
Secondary correlative evidence of anti-tumor response | Screening pre-treatment specimen Day - 8 through day -1; post treatment specimen Day 16-18
  As captured with tumoral Ki-67 and caspase staining on pre- and post-treatment specimens.
Secondary correlative evidence of disease control | baseline; 14-30 days prior to surgery, 30 and 90 days post resection surgery
  As measured by the HPV ctDNA with the NavDx assay
Occurrence of toxicity | Time of 1st treatment to 30 days post
  Adverse Events occurrence (Common Toxicity Criteria for Adverse Events), Immune-related adverse events of special interest, and hyperprogression will be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burtness, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Result] Smith TW, Aberger EW, Follick MJ, Ahern DK. Cognitive distortion and psychological distress in chronic low back pain. J Consult Clin Psychol. 1986 Aug;54(4):573-5. doi: 10.1037//0022-006x.54.4.573. No abstract available. PMID 2943767
- [Result] Rosol Z. [Etiology and propagation of myocardial irritation]. Cas Lek Cesk. 1971 Jul 23;110(30):717. No abstract available. Czech. PMID 5564292
- [Result] Cohen EEW, Soulieres D, Le Tourneau C, Dinis J, Licitra L, Ahn MJ, Soria A, Machiels JP, Mach N, Mehra R, Burtness B, Zhang P, Cheng J, Swaby RF, Harrington KJ; KEYNOTE-040 investigators. Pembrolizumab versus methotrexate, docetaxel, or cetuximab for recurrent or metastatic head-and-neck squamous cell carcinoma (KEYNOTE-040): a randomised, open-label, phase 3 study. Lancet. 2019 Jan 12;393(10167):156-167. doi: 10.1016/S0140-6736(18)31999-8. Epub 2018 Nov 30. PMID 30509740
- [Result] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Result] Vos JL, Elbers JBW, Krijgsman O, Traets JJH, Qiao X, van der Leun AM, Lubeck Y, Seignette IM, Smit LA, Willems SM, van den Brekel MWM, Dirven R, Baris Karakullukcu M, Karssemakers L, Klop WMC, Lohuis PJFM, Schreuder WH, Smeele LE, van der Velden LA, Bing Tan I, Onderwater S, Jasperse B, Vogel WV, Al-Mamgani A, Keijser A, van der Noort V, Broeks A, Hooijberg E, Peeper DS, Schumacher TN, Blank CU, de Boer JP, Haanen JBAG, Zuur CL. Neoadjuvant immunotherapy with nivolumab and ipilimumab induces major pathological responses in patients with head and neck squamous cell carcinoma. Nat Commun. 2021 Dec 22;12(1):7348. doi: 10.1038/s41467-021-26472-9. PMID 34937871
- [Result] Stewart RW. Cardiac transplantation at the Cleveland Clinic Foundation--the first 10 years. Clin Transpl. 1994:127-31. PMID 7547532
- [Result] Eklund AE, Eriksson G, Kallings LO, Liden S, Zetterquist S. [Venous leg ulcer, diagnosis and treatment]. Lakartidningen. 1980 Oct 1;77(40):3495-504. No abstract available. Swedish. PMID 7453348
- [Result] Bernstein RK. R-R interval studies: a simple office protocol for evaluation of autonomic neuropathy. Diabetes Care. 1984 Sep-Oct;7(5):510-3. doi: 10.2337/diacare.7.5.510b. No abstract available. PMID 6499643
- [Result] Gemzell C, Carlborl, Johansson ED, Roos P. Treatment of primary amenorrhoea with human pituitary and chorionic gonadotrophins. J Obstet Gynaecol Br Commonw. 1970 Jan;77(1):58-64. doi: 10.1111/j.1471-0528.1970.tb03408.x. No abstract available. PMID 5419871
- [Result] Albro PW, Fishbein L. Determination of prostaglandins by gas-liquid chromatography. J Chromatogr. 1969 Nov 11;44(3):443-51. doi: 10.1016/s0021-9673(01)92568-3. No abstract available. PMID 4311405
- [Result] Biktasova A, Hajek M, Sewell A, Gary C, Bellinger G, Deshpande HA, Bhatia A, Burtness B, Judson B, Mehra S, Yarbrough WG, Issaeva N. Demethylation Therapy as a Targeted Treatment for Human Papillomavirus-Associated Head and Neck Cancer. Clin Cancer Res. 2017 Dec 1;23(23):7276-7287. doi: 10.1158/1078-0432.CCR-17-1438. Epub 2017 Sep 15. PMID 28916527
- [Result] Kirst HA, Creemer LC, Paschal JW, Preston DA, Alborn WE Jr, Counter FT, Amos JG, Clemens RL, Sullivan KA, Greene JM. Antimicrobial characterization and interrelationships of dirithromycin and epidirithromycin. Antimicrob Agents Chemother. 1995 Jul;39(7):1436-41. doi: 10.1128/AAC.39.7.1436. PMID 7492081
- [Result] Davidovskii LIa. [Deficiency and transmembrane transport of water in pneumonia in young children]. Pediatriia. 1984 Mar;(3):54-5. No abstract available. Russian. PMID 6718162
- [Result] Glimelius B, Lahn M. Window-of-opportunity trials to evaluate clinical activity of new molecular entities in oncology. Ann Oncol. 2011 Aug;22(8):1717-25. doi: 10.1093/annonc/mdq622. Epub 2011 Jan 13. PMID 21239400
- [Result] Voillemin. [Urinary problems of paraplegics]. Rev Infirm. 1984 May;34(9):33-8. No abstract available. French. PMID 6564676
- [Result] Levy BP, Giaccone G, Besse B, Felip E, Garassino MC, Domine Gomez M, Garrido P, Piperdi B, Ponce-Aix S, Menezes D, MacBeth KJ, Risueno A, Slepetis R, Wu X, Fandi A, Paz-Ares L. Randomised phase 2 study of pembrolizumab plus CC-486 versus pembrolizumab plus placebo in patients with previously treated advanced non-small cell lung cancer. Eur J Cancer. 2019 Feb;108:120-128. doi: 10.1016/j.ejca.2018.11.028. Epub 2019 Jan 14. PMID 30654297
- [Result] Shapovalov AI, Shiriaev BI. [Synaptic interaction of individual motor neurons of the isolated frog spinal cord]. Neirofiziologiia. 1984;16(5):619-30. Russian. PMID 6096736
- [Result] Stansfeld CE, Wallis DI. Generation of an unusual depolarizing response in rabbit primary afferent neurones in the absence of divalent cations. J Physiol. 1984 Jul;352:49-72. doi: 10.1113/jphysiol.1984.sp015277. PMID 6086912
- [Result] Dendinger S, Brill WJ. Effect of the proline analogue baikiain on proline metabolism in Salmonella typhimurium. J Bacteriol. 1972 Dec;112(3):1134-41. doi: 10.1128/jb.112.3.1134-1141.1972. PMID 4565530